CLINICAL TRIAL: NCT00521872
Title: Stapled Trans Anal Rectal Resection (STARR) for Outlet Obstruction: Functional and Morphological Outcome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 33-2006
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2007-08

CONDITIONS: Surgery; Constipation
Keywords: surgery (STARR operation)
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: STARR Operation

SUMMARY:
This study compares pre- and postoperative (at 6 month) quality of life and pathomorphology of the pelvis (by MRI defecation) after a STARR procedure for outlet obstruction.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* All patients at our institution treated with the STARR operation

Exclusion criteria:

* Age under 18,
* Chronic or acute inflammatory disease of the bowel or rectum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pathomorphological changes of the pelvis (by MRI): intussuception, rectocele, defecation angles

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- UniversitätsSpital Zürich, Zurich, Switzerland